CLINICAL TRIAL: NCT07124000
Title: Effectiveness of T-DXd Across HER2-positive Solid Tumors in Patients Who Have Received Prior Systemic Treatment and Have no Satisfactory Alternative Treatment Options: A Hybrid Observational Study
Brief Title: DESTINY-PANTUMOUR04
Acronym: DP-04
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D781WR00001
Record Dates: First submitted 2025-08-13; First posted 2025-08-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Adenocarcinoma (NOS); Anal Cancer; Bladder Cancer; Cervical Cancer; Endometrial Cancer; Esophageal Cancer; Gall Bladder Cancer; Gastrointestinal Stromal Tumour; Head and Neck Cancer; Liver Cancer; Melanoma; Mouth Cancer; Nasopharangeal Cancer; Neuroendocrine, Gastrointestinal Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Renal Cell Carcinoma; Salivary Gland Cancer; Sarcoma; Small Cell Lung Cancer; Testicular Cancer; Throat Cancer; Thyroid Cancer; Urethral Cancer; Vaginal Cancer; Vulvar Cancer
MeSH Terms: conditions — Adenocarcinoma; Anus Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Gallbladder Neoplasms; Gastrointestinal Stromal Tumors; Head and Neck Neoplasms; Liver Neoplasms; Melanoma; Mouth Neoplasms; Gastrointestinal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell; Salivary Gland Neoplasms; Sarcoma; Small Cell Lung Carcinoma; Testicular Neoplasms; Thyroid Neoplasms; Urethral Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trastuzumab deruxtecan: Patients with locally advanced, unresectable, or metastatic HER-2 positive (IHC3+) solid tumours for whom a clinician decision has been made for treatment with T-DXd as part of routine clinical practice and in line with the FDA label
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan monotherapy
  Other Names: Enhertu

SUMMARY:
This study will evaluate the effectiveness of T-DXd in patients with HER2-positive (IHC 3+) locally advanced, unresectable, or metastatic solid tumors who have received prior systemic treatment for metastatic or advanced disease and have no satisfactory alternative treatment options in a real-world setting in the US

DETAILED DESCRIPTION:
This study is a multicenter, hybrid, observational study of approximately 100 prospectively enrolled patients with HER2-positive (IHC 3+) solid tumors in the US initiated on trastuzumab deruxtecan (T-DXd) as per FDA label in routine clinical practice and enrolled at the point of starting treatment with T-DXd. Patients with locally advanced, unresectable, or metastatic HER2-positive (IHC 3+) solid tumors who have received prior systemic treatment for metastatic or advanced disease and have no satisfactory alternative treatment options will be eligible for inclusion. Patients with breast, colorectal, non-small cell lung cancer (NSCLC), gastric/gastroesophageal junction (GEJ) cancers, and haematological malignancies are not eligible for this study.

Approximately 30 sites will be selected including community oncology practices, hospital systems and academic medical centers (AMCs), with a focus on enrolling a patient population representative of real-world care with the majority of patients from community settings. The primary objective of the study is to assess real world response rate and real world duration of response, and the secondary objective is to assess real world time to treatment discontinuation and real world time to next treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years
2. Patients with locally advanced, unresectable, or metastatic HER2-positive (IHC 3+) solid tumors who have received prior systemic treatment for metastatic or advanced disease and have no satisfactory alternative treatment options as determined by the Investigator (see Exclusion Criterion 1 for excluded solid tumors);
3. A clinician decision has been made for treatment with T-DXd in accordance with the FDA label;
4. HER2-positive (IHC 3+) by local testing prior to study enrolment at the time of signed and dated informed consent;
5. Patients who are willing and able to provide a signed and dated informed consent.

Exclusion Criteria:

1. Primary diagnosis of adenocarcinoma of the breast, adenocarcinoma of the colon or rectum, NSCLC, adenocarcinoma of the gastric body or gastroesophageal junction or hematological malignancies;
2. Prior T-DXd therapy;
3. Patients without a baseline assessment of tumor burden undertaken prior to initiating T-DXd.
4. Patient is participating in a clinical trial at time of enrolment

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients for whom a clinician decision has been made for treatment with T-DXd as part of routine clinical practice and in line with the FDA label, but who have not yet started therapy with T-DXd
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Real world response rate (rwRR) | Through study completion, up to 2.5 years after enrolment
  rwRR is defined as the proportion of patients with a clinician assessment of complete or partial response while on T-DXd treatment
Real world duration of response (rwDoR) | Through study completion, up to 2.5 years after enrolment
  rwDoR is defined as the time from first physician reported complete or partial response until time of progression or death

SECONDARY OUTCOMES:
Real world time to treatment discontinuation (rwTTD) | Through study completion, up to 2.5 years after enrolment
  rwTTD is defined as the time from first administration of T-DXd to the date of the clinican decision to discontinue treatment with T-DXd or patient death while on T-DXd therapy
Real world time to next treatment (rwTTNT) | Through study completion, up to 2.5 years after enrolment
  rwTTNT is defined as the time from the date of first administration of T-DXd to the date of first administration of the next line of treatment or death

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Research Site, Birmingham, Alabama
  - Research Site, Casa Grande, Arizona
  - Research Site, Coral Springs, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, O'Fallon, Illinois
  - Research Site, Wilson, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Maumee, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/